CLINICAL TRIAL: NCT05098587
Title: Are Changes in Pain Perception Associated With Changes in Brain Activity Patterns in Persons With Spinal Cord Injury and Neuropathic Pain After a Virtual Walking Training Program - A Pilot Study
Brief Title: Brain Activity Patterns in Persons With Spinal Cord Injury and Neuropathic Pain After a Virtual Walking Training Program
Acronym: VRandMRI
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Haute Ecole de Santé Vaud (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-13
Record Dates: First submitted 2021-09-13; First posted 2021-10-28 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
Keywords: functional magnetic resonance imaging; brain activity patterns
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this pilot study is to explore the association of changes in pain perception with changes in brain activity (functional Magnetic Resonance Imaging (fMRI)) and metabolic (Magnetic Resonance Spectroscopy (MRS)) patterns of individuals with SCI and chronic NeP after a Virtual Walk (VW) therapy. The brain activity patterns will be assessed in resting state and under a specific task, before and after a VW training program, done as part of the clinical routine, as well as at a four weeks follow-up.

The results of this pilot study will serve as basis for a bigger project that aims to investigate and compare brain activity and long-term effects of non-immersive VW therapy on chronic NeP in individuals with SCI (traumatic SCI with chronic NeP at- or below level, complete or incomplete) taking into account confounding factors such as time since injury, level of injury and type of NeP.

DETAILED DESCRIPTION:
This pilot study consists of specific assessments at four different time points (T0=screening, T1=baseline, pre measurement, T2=post measurement, T3=four week follow-up).

The physiotherapeutical assessment at T0 involves the evaluation of the imagery capacity. At T1, the participant will be assessed for baseline measures before starting with the VW training. At T2 (after the last VW training) and at T3 (four weeks after the last VW training), the participant will be assessed for outcome measures.

Sociodemographic and clinical characteristics (age, sex, education level, workability, age at injury, lesion level, comorbidities, complications, concomitant injuries, SCI pain basic dataset 2.0 and medication) will be collected in the screening/recruitment phase but only used after receiving informed consent from each participant.

Participants will undergo a non-invasively MRI examination without application of contrast agents. The functional activity of the brain will be assessed by a blood oxygenation level-dependent (BOLD) fMRI. The metabolic profile will be assessed non-invasively by means of single voxel MRS. Prior to the fMRI and MRS measurements, a high-resolution anatomical MRI will be performed, which serves for tissue segmentation and planning purposes.

The MRI will consist out of the following sequences conducted in an MRI scanner (six minutes duration each):

1. MRS sequence: The metabolic profile will be assessed with single voxel spectroscopy in the Anterior Cingulate Cortex and the Thalamus.
2. Resting-state fMRI: The participant will stay rested with open eyes and does not have to perform a specific task.
3. Task-based fMRI: In an on-off scheme, a sequence of neutral (not pain related) pictures on a screen, mounted outside of the MRI machine will be shown. The pictures will change every 20 seconds in a random order to keep the participant alert.
4. Task-based fMRI: In an on-off scheme, a sequence of pain-related pictures on a screen, mounted outside of the MRI machine will be shown. The pictures will change every 20 seconds in a random order to keep the participant alert.
5. Resting-state fMRI: The participant will stay rested with open eyes and does not have to execute a task.

The pain images shown during the task-based fMRI are a validated set of pictures.

The participants will receive a pain diary. This pain diary is filled in daily for the one-week period before the baseline assessments, during the VW therapy and in the week before the last assessments at T3. To minimise the risk of missing data in the pain diary the participants will be called one week before T3 and get reminded to fill in the pain diary.

Before starting with the VW therapy the participants will first perform a subitem of the standardised Graded Motor Imagery (GMI) training over four weeks, five times a day using the Recognise Foot App and the Recognise Hand App. The participants will train their capacity to perform a left-right discrimination for hands and feet. This training will help to improve the therapeutic effect of the following VW therapy program, by improving the imagery capacity. Reaction time as well as accuracy while performing a left-right discrimination task will be measured. More than 80% correct answers and a reaction time of less than two seconds is interpreted as good imagery capacity. The imagery capacity will be assessed right before the start of the discrimination training, after two weeks and after four weeks. This serves on one hand as information about participant characteristics and on the other hand as a control mechanism that each participant keeps performing this training.

After the discrimination training, the participants will perform a non-immersive VW therapy program at the pain clinic, which consists of five sessions of 10 to 20 minutes per week, over a two-week period, then three treatments per week for the following two weeks and finally in the last two weeks only two treatments per week are scheduled. This is the standard protocol for this kind of therapy and is not changed in any way for the participants of the MRI study. For the VW, the participants will sit on an electric wheelchair in front of a canvas with an integrated camera. The camera films the participant's head and trunk, which are then projected on the canvas, overlapping with the recording of the feet of an actor walking. This way the participants will see themselves walk through a forest from a third-person view. To improve the embodiment, the participants will be asked to swing their arms in the rhythm of the gait and imagine that they are walking themselves through the forest. In addition to this, the chair moves minimally in the frontal plane to imitate the natural movements of the pelvis while walking.

ELIGIBILITY:
Inclusion Criteria:

* Passed neurological, physiotherapeutic and psychological assessments and team decision to take part on VW
* Age ≧ 18
* Traumatic SCI (> 1 year) confirmed by MRI or CT
* Neuropathic at or below level spinal cord injury pain for at least 3 months diagnosed by a neurologist following the CanPain Clinical Practice Guidelines and ISCIP classification
* Good German skills (understand questionnaires and instructions)
* Ability to draw with a pen
* Ability to swing the arms

Exclusion Criteria:

* Claustrophobia
* Non-acceptance of the paraplegia
* Psychiatric disorders
* Epilepsy
* Other neurological, psycho-logical or cognitive impairments
* Pregnancy
* Spasticity that would interfere with MRI
* Extensive dose of opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twelve individuals with SCI and NeP will be recruited at the Centre for Pain Medicine, Swiss Paraplegic Centre, Nottwil. A neurologist will check for inclusion and exclusion criteria.
  Patients, who will be screened routineously as part of the ordinary clinical visit by a neurologist, a physiotherapist and a psychologist for their eligibility to take part in the clinical VW program, will additionally be screened for their participation in the intended study. These assessments include checking inclusion and exclusion criteria and a diagnosis using the SCI pain basic dataset 2.0.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Change of N-Acetyl-Aspartate in the anterior cingulate cortex | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Non-invasive MRI-based metabolic marker measured under various conditions (resting state, painful images, non-painful images)

SECONDARY OUTCOMES:
Change of Choline | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Non-invasive MRI-based metabolic marker (resting state, painful images, non-painful images)
Alteration of Creatine | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Non-invasive MRI-based metabolic marker
Alteration of myo-Inositol | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Non-invasive MRI-based metabolic marker
BOLD signal changes during task-based and resting state functional MRI | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Task-based and resting state functional MRI sequences are applied and BOLD signal changes are examined. A whole-brain and seed-based connectivity analysis are used and linked to pain processing and perception.
Pain diary | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  A pain diary using the numeric pain rating scale from 0 = "no pain at all" to 10 = "worst imaginable pain", to assess pain intensity during the course of the study and in follow-up.
Pain description list | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire containing 12 descriptions of pain to assess the quality of pain (how the pain is perceived) Patients have to rate each description on a scale ranging from 0 = "completely disagree" to 3 = "fully agree" Items 1 to 8 are only descriptively evaluated. The sum of items 9 to 12 is the affective score whereas a high value is indicating a high affective burden and a low value is equal to a low affective burden.
Chronic pain grading scale | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire to assess the severity of chronic pain and its impact on daily activities containing 7 items that must be rated on a NRS ranging from 0 = "no pain", "no limitation"; to 10 = "worst imaginable pain"/limitation". Higher values thus indicating more pain/limitation.
The Marburg questionnaire on habitual health findings | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire to assess general wellbeing containing 7 items that have to be rated on a rating scale ranging from 0 = "completely disagree" to 5 = "completely agree". A high score in this questionnaire indicates high well-being.
WHO-QoL-BREF | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire containing 26 items to assess quality of life rated on a rating scale ranging from 1 = "very bad"/"very unhappy"/"not at all"/"never" to 5 = "very good"/"very happy"/"absolutely"/"always". Depending on the statements the scores have to be inversed to calculate the score. Higher scores indicate better quality of life. There are four domain scores that result from this questionnaire: physical domain, psychological domain, social relationships domain and environment domain.
Pain catastrophizing scale | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire containing 13 items/statements to assess pain catastrophizing on a rating scale ranging from 0 = "never true" to 4 = "always true". A high score indicates a high degree of pain catastrophizing.
Questions about pain chronification | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire to assess pain chronification consisting of ten questions. The single questions help to classify the stadium of pain chronification ranging from stadium I = mild chronification to stadium III = heavy chronification.
SCI independence measure III - self-reported version | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire addressing the functional impairment including 17 items assessing the grade of necessary aid versus ability to do it on their own for specific daily activities with ratings ranging from 0 = "not able to do a task" to 8 = "no or minimal aid". The higher the score the more independent the person.
Depression, Anxiety & Stress Scale | Three measurement time points: Baseline (T1), six weeks after baseline (T2), ten weeks after after baseline (T3)
  Questionnaire to assess depression, anxiety and stress using 21 items rated on a scale from 0 = "absolutely disagree" or "never" to 3 = "strong agreement" or "most of the time". Because the items are negatively formulated a high score indicates a high grade of depression, anxiety or stress. Each domain score consists of 7 items.
Patient Global Impression of Change | Two measurement time points: only T2 (six weeks after baseline) and T3 (ten weeks after baseline))
  One question to assess the subjective global impression of change after the therapy. The choice options range from "very much better than before" to "very much worse than before" with "unchanged" as the middle/neutral value.

OTHER OUTCOMES:
Sociodemographic and clinical characteristics | At the beginning and at follow up.
  Collected during clinical routine: age, sex, pain duration, age at injury, lesion level, comorbidities, concomitant injuries, pain severity, pain distribution and quality, medication, education level, workability, functional impairment, motor imagery capacity and habits like smoking, quantity of alcohol or caffeine-containing potables.

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre; Centre for pain medicine, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryce TN, Ragnarsson KT. Pain after spinal cord injury. Phys Med Rehabil Clin N Am. 2000 Feb;11(1):157-68. PMID 10680163
- [Background] Fekete C, Eriks-Hoogland I, Baumberger M, Catz A, Itzkovich M, Luthi H, Post MW, von Elm E, Wyss A, Brinkhof MW. Development and validation of a self-report version of the Spinal Cord Independence Measure (SCIM III). Spinal Cord. 2013 Jan;51(1):40-7. doi: 10.1038/sc.2012.87. Epub 2012 Aug 14. PMID 22890418
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Background] Guy SD, Mehta S, Casalino A, Cote I, Kras-Dupuis A, Moulin DE, Parrent AG, Potter P, Short C, Teasell R, Bradbury CL, Bryce TN, Craven BC, Finnerup NB, Harvey D, Hitzig SL, Lau B, Middleton JW, O'Connell C, Orenczuk S, Siddall PJ, Townson A, Truchon C, Widerstrom-Noga E, Wolfe D, Loh E. The CanPain SCI Clinical Practice Guidelines for Rehabilitation Management of Neuropathic Pain after Spinal Cord: Recommendations for treatment. Spinal Cord. 2016 Aug;54 Suppl 1:S14-23. doi: 10.1038/sc.2016.90. PMID 27444715
- [Background] Jackson PL, Meltzoff AN, Decety J. How do we perceive the pain of others? A window into the neural processes involved in empathy. Neuroimage. 2005 Feb 1;24(3):771-9. doi: 10.1016/j.neuroimage.2004.09.006. PMID 15652312
- [Background] Klasen BW, Hallner D, Schaub C, Willburger R, Hasenbring M. Validation and reliability of the German version of the Chronic Pain Grade questionnaire in primary care back pain patients. Psychosoc Med. 2004 Oct 14;1:Doc07. PMID 19742049
- [Background] Kleinloog D, Rombouts S, Zoethout R, Klumpers L, Niesters M, Khalili-Mahani N, Dahan A, van Gerven J. Subjective Effects of Ethanol, Morphine, Delta(9)-Tetrahydrocannabinol, and Ketamine Following a Pharmacological Challenge Are Related to Functional Brain Connectivity. Brain Connect. 2015 Dec;5(10):641-8. doi: 10.1089/brain.2014.0314. Epub 2015 Sep 21. PMID 26390148
- [Background] Mehta S, Guy SD, Bryce TN, Craven BC, Finnerup NB, Hitzig SL, Orenczuk S, Siddall PJ, Widerstrom-Noga E, Casalino A, Cote I, Harvey D, Kras-Dupuis A, Lau B, Middleton JW, Moulin DE, O'Connell C, Parrent AG, Potter P, Short C, Teasell R, Townson A, Truchon C, Wolfe D, Bradbury CL, Loh E. The CanPain SCI Clinical Practice Guidelines for Rehabilitation Management of Neuropathic Pain after Spinal Cord: screening and diagnosis recommendations. Spinal Cord. 2016 Aug;54 Suppl 1:S7-S13. doi: 10.1038/sc.2016.89. PMID 27444717
- [Background] Meyer K, Sprott H, Mannion AF. Cross-cultural adaptation, reliability, and validity of the German version of the Pain Catastrophizing Scale. J Psychosom Res. 2008 May;64(5):469-78. doi: 10.1016/j.jpsychores.2007.12.004. PMID 18440399
- [Background] Reckziegel D, Vachon-Presseau E, Petre B, Schnitzer TJ, Baliki MN, Apkarian AV. Deconstructing biomarkers for chronic pain: context- and hypothesis-dependent biomarker types in relation to chronic pain. Pain. 2019 May;160 Suppl 1(Suppl 1):S37-S48. doi: 10.1097/j.pain.0000000000001529. PMID 31008848
- [Background] Siddall PJ, McClelland JM, Rutkowski SB, Cousins MJ. A longitudinal study of the prevalence and characteristics of pain in the first 5 years following spinal cord injury. Pain. 2003 Jun;103(3):249-257. doi: 10.1016/S0304-3959(02)00452-9. PMID 12791431
- [Background] Turk DC, Dworkin RH, Allen RR, Bellamy N, Brandenburg N, Carr DB, Cleeland C, Dionne R, Farrar JT, Galer BS, Hewitt DJ, Jadad AR, Katz NP, Kramer LD, Manning DC, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robinson JP, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Witter J. Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. Pain. 2003 Dec;106(3):337-345. doi: 10.1016/j.pain.2003.08.001. PMID 14659516
- [Background] Upadhyay J, Maleki N, Potter J, Elman I, Rudrauf D, Knudsen J, Wallin D, Pendse G, McDonald L, Griffin M, Anderson J, Nutile L, Renshaw P, Weiss R, Becerra L, Borsook D. Alterations in brain structure and functional connectivity in prescription opioid-dependent patients. Brain. 2010 Jul;133(Pt 7):2098-114. doi: 10.1093/brain/awq138. Epub 2010 Jun 16. PMID 20558415
- [Background] Widerstrom-Noga E, Biering-Sorensen F, Bryce TN, Cardenas DD, Finnerup NB, Jensen MP, Richards JS, Siddall PJ. The International Spinal Cord Injury Pain Basic Data Set (version 2.0). Spinal Cord. 2014 Apr;52(4):282-6. doi: 10.1038/sc.2014.4. Epub 2014 Jan 28. PMID 24469147
- [Background] Whitfield-Gabrieli S, Nieto-Castanon A. Conn: a functional connectivity toolbox for correlated and anticorrelated brain networks. Brain Connect. 2012;2(3):125-41. doi: 10.1089/brain.2012.0073. Epub 2012 Jul 19. PMID 22642651
- [Result] Austin PD, Siddall PJ. Virtual reality for the treatment of neuropathic pain in people with spinal cord injuries: A scoping review. J Spinal Cord Med. 2021 Jan;44(1):8-18. doi: 10.1080/10790268.2019.1575554. Epub 2019 Feb 1. PMID 30707649
- [Result] Chi B, Chau B, Yeo E, Ta P. Virtual reality for spinal cord injury-associated neuropathic pain: Systematic review. Ann Phys Rehabil Med. 2019 Jan;62(1):49-57. doi: 10.1016/j.rehab.2018.09.006. Epub 2018 Oct 9. PMID 30312665
- [Result] de Araujo AVL, Neiva JFO, Monteiro CBM, Magalhaes FH. Efficacy of Virtual Reality Rehabilitation after Spinal Cord Injury: A Systematic Review. Biomed Res Int. 2019 Nov 13;2019:7106951. doi: 10.1155/2019/7106951. eCollection 2019. PMID 31828120
- [Result] Duncan NW, Northoff G. Overview of potential procedural and participant-related confounds for neuroimaging of the resting state. J Psychiatry Neurosci. 2013 Mar;38(2):84-96. doi: 10.1503/jpn.120059. PMID 22964258
- [Result] Eick J, Richardson EJ. Cortical activation during visual illusory walking in persons with spinal cord injury: a pilot study. Arch Phys Med Rehabil. 2015 Apr;96(4):750-3. doi: 10.1016/j.apmr.2014.10.020. Epub 2014 Nov 15. PMID 25461820
- [Result] Mahnig S, Landmann G, Stockinger L, Opsommer E. Pain assessment according to the International Spinal Cord Injury Pain classification in patients with spinal cord injury referred to a multidisciplinary pain center. Spinal Cord. 2016 Oct;54(10):809-815. doi: 10.1038/sc.2015.219. Epub 2016 Jan 12. PMID 26754471
- [Result] Moseley LG. Using visual illusion to reduce at-level neuropathic pain in paraplegia. Pain. 2007 Aug;130(3):294-298. doi: 10.1016/j.pain.2007.01.007. Epub 2007 Mar 1. PMID 17335974
- [Result] Moseley GL, Flor H. Targeting cortical representations in the treatment of chronic pain: a review. Neurorehabil Neural Repair. 2012 Jul-Aug;26(6):646-52. doi: 10.1177/1545968311433209. Epub 2012 Feb 13. PMID 22331213
- [Result] Opsommer E, Chevalley O, Korogod N. Motor imagery for pain and motor function after spinal cord injury: a systematic review. Spinal Cord. 2020 Mar;58(3):262-274. doi: 10.1038/s41393-019-0390-1. Epub 2019 Dec 13. PMID 31836873
- [Result] Pattany PM, Yezierski RP, Widerstrom-Noga EG, Bowen BC, Martinez-Arizala A, Garcia BR, Quencer RM. Proton magnetic resonance spectroscopy of the thalamus in patients with chronic neuropathic pain after spinal cord injury. AJNR Am J Neuroradiol. 2002 Jun-Jul;23(6):901-5. PMID 12063213
- [Result] Richardson EJ, McKinley EC, Rahman AKMF, Klebine P, Redden DT, Richards JS. Effects of virtual walking on spinal cord injury-related neuropathic pain: A randomized, controlled trial. Rehabil Psychol. 2019 Feb;64(1):13-24. doi: 10.1037/rep0000246. Epub 2018 Nov 8. PMID 30407030
- [Result] Soler MD, Kumru H, Pelayo R, Vidal J, Tormos JM, Fregni F, Navarro X, Pascual-Leone A. Effectiveness of transcranial direct current stimulation and visual illusion on neuropathic pain in spinal cord injury. Brain. 2010 Sep;133(9):2565-77. doi: 10.1093/brain/awq184. Epub 2010 Aug 4. PMID 20685806
- [Result] Widerstrom-Noga E, Pattany PM, Cruz-Almeida Y, Felix ER, Perez S, Cardenas DD, Martinez-Arizala A. Metabolite concentrations in the anterior cingulate cortex predict high neuropathic pain impact after spinal cord injury. Pain. 2013 Feb;154(2):204-212. doi: 10.1016/j.pain.2012.07.022. Epub 2012 Nov 8. PMID 23141478
- [Result] Widerstrom-Noga E, Cruz-Almeida Y, Felix ER, Pattany PM. Somatosensory phenotype is associated with thalamic metabolites and pain intensity after spinal cord injury. Pain. 2015 Jan;156(1):166-174. doi: 10.1016/j.pain.0000000000000019. PMID 25599312
- [Result] Wrigley PJ, Press SR, Gustin SM, Macefield VG, Gandevia SC, Cousins MJ, Middleton JW, Henderson LA, Siddall PJ. Neuropathic pain and primary somatosensory cortex reorganization following spinal cord injury. Pain. 2009 Jan;141(1-2):52-9. doi: 10.1016/j.pain.2008.10.007. Epub 2008 Nov 21. PMID 19027233
- See also: Declaration of Helsinki — https://www.wma.net/what-we-do/medical-ethics/declaration-of-helsinki/
- See also: Ordinance on Human Research with the Exception of Clinical trials (HRO), swiss law — https://www.admin.ch/opc/en/classified-compilation/20121177/index.html
- See also: Human Research Act (HRA), swiss law — http://www.admin.ch/opc/en/classified-compilation/20121176/201401010000/810.305.pdf